CLINICAL TRIAL: NCT02339298
Title: Impact of Intraoperative Music Application on Postoperative Behaviour in Children and Adolescents.
Brief Title: Intraoperative Music Application and Postoperative Behaviour in Children and Adolescents.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Children's Hospital, Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Music study StV 10/09
Record Dates: First submitted 2014-12-12; First posted 2015-01-15 (Estimated); Last update posted 2015-11-10 (Estimated); Status verified 2015-11

CONDITIONS: Postoperative Behaviour
Keywords: Music Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Music group (Active Comparator): music application
  Interventions: Other: music application; Drug: a caudal block
- Control group (Sham Comparator): only headphones
  Interventions: Other: only headphones; Drug: a caudal block

INTERVENTIONS:
Other: music application — music is applied during anaesthesia using headphones
  Arms: Music group
Other: only headphones — music is not applied, only headphones are placed
  Arms: Control group
Drug: a caudal block

SUMMARY:
The purpose of the study is to evaluate whether intraoperative music application has a positive impact on postoperative behavior in children and adolescents.

DETAILED DESCRIPTION:
After induction of anesthesia, paralyzation of the patient and subsequent intubation, a caudal block is applied. After positioning of the patient, headphones are placed on the patients head and in case of the interventional group, music is played. Previously, the volume of the music is adjusted to a range from 50 to 60 decibel. Headphones are removed before extubation.

Postoperative behaviour is evaluated by parents and by caretaking personnel in the recovery room at arrival, after 15 minutes and before discharge to the ward and at home by parents after one, two and four weeks using questionnaires.

sample size calculation: n = minimal number of required probands π = 70% (proportion of interest) → 0.7 π0 = 50% (null hypothesis proportion) → 0.5 μ = (100% - 90%power) → 1.28 v = 1.96 (level of significance p=0.05)

n > [ μ√ π(1- π) + v√ π0(1- π0)]2 / (π - π0) n > 61.4 + correction for drop-outs (+10%) n = 70 per group → 140 probands in total

ELIGIBILITY:
Inclusion Criteria:

* age: 4-16 years
* American Society of Anesthesiologists (ASA) physical status of 1 and 2
* elective inguinal herniotomy or circumcision
* general anaesthesia with sevoflurane and caudal block
* written informed consent available

Exclusion Criteria:

* age <4 or >16.99 years
* ASA physical status of 3 or higher
* emergency surgery
* no general anaesthesia with sevoflurane or/and caudal block
* no written informed consent available

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 140 (Actual)
Dates: Start 2009-07; Primary Completion 2015-10 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Occuring of a behaviour change | patients are followed during the first 4 weeks after the operation
  Patients are followed during the first 4 weeks after the operation by parents using a questionnaire in order to detect behaviour changes after the operation.

SECONDARY OUTCOMES:
occurring of postoperative vomiting | baseline
occurring of postoperative vomiting | 15 min after arrival at the recovery room
occurring of postoperative vomiting | before discharge to the ward, which means after an expected average stay of 2 hours at the recovery room
rating of the behaviour of the child in the recovery room by parents using a questionnaire | baseline
rating of the behaviour of the child in the recovery room by parents using a questionnaire | 15 min after arrival at the recovery room
rating of the behaviour of the child in the recovery room by parents using a questionnaire | before discharge to the ward, which means after an expected average stay of 2 hours at the recovery room
rating of the behaviour of the child in the recovery room by caretaking personnel using a questionnaire | baseline
rating of the behaviour of the child in the recovery room by caretaking personnel using a questionnaire | 15 min after arrival at the recovery room
rating of the behaviour of the child in the recovery room by caretaking personnel using a questionnaire | before discharge to the ward, which means after an expected average stay of 2 hours at the recovery room

CONTACTS AND LOCATIONS:
Overall Officials: Markus Weiss, Prof., Principal Investigator — University Children's Hospital, Zurich
Locations (1):
- University Children's Hospital, Zurich, Canton of Zurich, Switzerland